CLINICAL TRIAL: NCT02537912
Title: Effects of Peanut Skin Extract on Blood Glucose Regulation and Body Fat Reduction
Brief Title: Blood Glucose and Body Fat Regulatory Effect of Peanut Skin Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, You-Cheng Shen, School of Health Diet and Industry Managment, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS13167
Record Dates: First submitted 2015-08-23; First posted 2015-09-02 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Obesity
Keywords: peanut skin; body fat; blood glucose; waistline; body weight
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugarlock® (Active Comparator): Subjects ingested 2 capsules Sugarlock® (Experimental group) in the morning and 2 capsules in the evening (4 capsules/d) for a total of 6 weeks.
  Interventions: Dietary Supplement: Sugarlock®
- Placebo (Placebo Comparator): Subjects ingested 2 capsules placebo (Control group) in the morning and 2 capsules in the evening (4 capsules/d) for a total of 6 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Sugarlock® — Subjects ingested 2 capsules (Experimental group) in the morning and 2 capsules in the evening (4 capsules/d) for a total of 6 weeks. Anthropometric measurements such as body weight, body fat, waistline, hipline, blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]) and blood biochemical parameters including FBG, albumin, TC, TG, HDL-C, LDL-C, Cr, BUN, AST and ALT were measured every three weeks. Five subjects were randomly selected to take MRI abdominal scans before and after the trial. After 6-week consumption, anthropometric measurements were examined on week 8 for a follow-up observation.
  Other Names: peanut skin
  Arms: Sugarlock®
Dietary Supplement: Placebo — Subjects ingested 2 capsules placebo in the morning and 2 capsules in the evening (4 capsules/d) for a total of 6 weeks. Anthropometric measurements such as body weight, body fat, waistline, hipline, blood pressure (systolic blood pressure [SBP] and diastolic blood pressure [DBP]) and blood biochemical parameters including FBG, albumin, TC, TG, HDL-C, LDL-C, Cr, BUN, AST and ALT were measured every three weeks. Five subjects were randomly selected to take MRI abdominal scans before and after the trial. After 6-week consumption, anthropometric measurements were examined on week 8 for a follow-up observation.
  Arms: Placebo

SUMMARY:
The regulatory effects of the peanut skin extract (Sugarlock®) on body fat and blood glucose was demonstrated in a double-blind, placebo-controlled study. .

DETAILED DESCRIPTION:
Peanut skins, a by-product of peanut processing industry, is usually discarded as a waste in despite of the high content of phenolic compounds. Polyphenol extract from peanut skins has been demonstrated to inhibit α-amylase activity in vitro. Hence, the aim of this study was to evaluate the regulatory effects of the peanut skin extract on blood glucose and body fat by a double-blind, placebo-controlled, clinical study. Subjects with simple obesity (body mass index [BMI] ≥ 27 or body fat ≥ 30%) ingested 4 Sugarlock® (n = 16) capsules or placebo (n = 14) a day for a total of 6 weeks. Anthropometric measurements (body weight, body fat, blood pressure) and blood biochemical markers including fasting blood glucose (FBG), albumin, total cholesterol (TC), triglyceride (TG), HDL-C, LDL-C, creatinine (Cr), blood urea nitrogen (BUN), AST, ALT were examined every three weeks. Also, 5 subjects were randomly selected for MRI scans to examine the distribution and thickness of abdominal fat layers before and after the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 20-70 years;
* Body mass index (BMI) ≥ 27 or body fat ≥ 30;
* No history of serious diseases associated with heart, liver, kidney, endocrine systems or other organs;
* No drugs consumption.

Exclusion Criteria:

* BMI >35;
* Alcoholic;
* US-controlled diabetics;
* Stoke in past one year;
* High blood pressure;
* Mental diseases or melancholia;
* Pregency or breast-feeding a child.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The changes of body fat of the subjects. | 6 weeks
  values change of body fat (%) between before to after 6 weeks

SECONDARY OUTCOMES:
The changes of fasting blood glucose (FBG) of the subjects | 6 weeks
  values change of fasting blood glucose (FBG) between before to after 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: You-Cheng Mr Shen, Ph.D., Principal Investigator — Chung Shan Medical University

REFERENCES:
- [Background] Grussu D, Stewart D, McDougall GJ. Berry polyphenols inhibit alpha-amylase in vitro: identifying active components in rowanberry and raspberry. J Agric Food Chem. 2011 Mar 23;59(6):2324-31. doi: 10.1021/jf1045359. Epub 2011 Feb 17. PMID 21329358
- [Background] McDougall GJ, Shpiro F, Dobson P, Smith P, Blake A, Stewart D. Different polyphenolic components of soft fruits inhibit alpha-amylase and alpha-glucosidase. J Agric Food Chem. 2005 Apr 6;53(7):2760-6. doi: 10.1021/jf0489926. PMID 15796622
- [Background] Yu Y, Gao F, Deng X, Pu X, Zhang M, Pang Y. Inhibitory effect of polyphenol extracts from peanut shells on the activity of pancreatic α-amylase activity in vitro. J Food Agric Environ. 2013; 11: 38-42.J Agric Food Chem. 2005; 53: 2760-2766.